CLINICAL TRIAL: NCT05435625
Title: Fractional Microneedling Radiofrequency Versus Fractional Carbon Dioxide Laser in Combination With Minoxidil for the Treatment of Androgenetic Alopecia
Brief Title: Fractional Laser Versus Radiofrequency in Androgenetic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Assistant Professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Laser-RF:AGA
Record Dates: First submitted 2022-03-11; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FCO2 (Active Comparator): Fractional Carbon dioxide laser
  Interventions: Procedure: FCO2
- FRF (Active Comparator): Fractional Microneedling Radiofrequency
  Interventions: Procedure: FRF

INTERVENTIONS:
Procedure: FCO2 — Fractional Carbon dioxide laser
  Arms: FCO2
Procedure: FRF — Fractional Microneedling Radiofrequency
  Arms: FRF

SUMMARY:
Patients with Androgenetic alopecia will be randomized into 2 groups; Group FCO2 receiving Fractional CO2 or Group FRF receiving Fractional Microneedling Radiofrequency.

DETAILED DESCRIPTION:
Group FCO2 will be to receiving fractional CO2 to one randomized side of the scalp, and Group FRF will be receiving Fractional Microneedling radiofrequency to one randomized side of the scalp.

All patients will receive 4 sessions with 4-week intervals.each session will be followed by immediate topical application of 6 puffs (=1 mL) of minoxidil 5% solution twice daily and also in between the sessions and during follow up period

ELIGIBILITY:
Inclusion Criteria:

* • both genders are included.

  * Patients above 18 years old.

Exclusion Criteria:

* • Patients with patchy hair loss.

  * Patients with Telogen Effluvium or diffuse alopecia areata.
  * Patients with cicatricial alopecias.
  * Patients with associated inflammatory scalp disorders such as psoriasis or seborrheic dermatitis.
  * Patients with collagen vascular disorders.
  * Prior use of topical steroids on scalp in the previous 2 weeks.
  * Prior use of systemic steroids in the previous 1 month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Global improvement Assessment | 6months-1 year
  Photographs will be taken with a Canon camera under controlled light in approximately the same position, taken at baseline, after 4 treatment sessions (16 weeks post treatment) and 2 months after follow-up (24 weeks post treatment). First clinical assessment will be performed based on the clinical change from baseline at 16 weeks post treatment. Change in the clinical will be measured on a 6 point scale; (-1) worsening, (0) no improvement, (1) less than 25% improvement, (2) 25-50% improvement, (3) 50-75% improvement, (4) more than 75% improvement. A higher numerical means a better outcome.
Clinical Global improvement Assessment | 6months-1 year
  Photographs will be taken with a Canon camera under controlled light in approximately the same position, taken at baseline, after 4 treatment sessions (16 weeks post treatment) and 2 months after follow-up (24 weeks post treatment). Second clinical assessment will be performed based on the clinical change from 16 weeks post treatment to 24 weeks post treatment. Change in the clinical will be measured on a 6 point scale; (-1) worsening, (0) no improvement, (1) less than 25% improvement, (2) 25-50% improvement, (3) 50-75% improvement, (4) more than 75% improvement. A higher numerical means a better outcome.
Phototrichogram assessment. | months-1 year
  A phototrichogram system (Dino-Lite; AnMo Electronics, Taiwan)will be used to evaluate the number of hairs. A higher numerical means a better outcome.
Phototrichogram assessment. | 2 months
  A phototrichogram system (Dino-Lite; AnMo Electronics, Taiwan)will be used to evaluate the thickness of hairs. A higher numerical means a better outcome.
Patient satisfaction | 6months-1 year
  Participants will be also asked to give their assessment on a scale of 4, (0) no satisfaction (1) slight satisfation, (2) moderate satisfaction, (3) marked satisfaction. A higher numerical means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy Hospital, Cairo, El Manial, Egypt